CLINICAL TRIAL: NCT05155514
Title: Comparison of the Relationship Between Preoperatively Measured Pulse Wave Velocity and Hemodynamic Changes During Anesthesia Induction in Hypertensive and Normotensive Patients.
Brief Title: Pulse Wave Velocity and Hemodynamic Response During Anesthesia Induction in Hypertensive Patients
Acronym: AS
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SİNAN YILMAZ, Associate Professor, Aydin Adnan Menderes University
Other Study IDs: Arterial stiffness
Record Dates: First submitted 2021-12-03; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Arterial Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group H: Hypertension group (Group H):
  * Patients with a previous diagnosis of hypertension
  * Patients receiving antihypertensive therapy
  * Systolic blood pressure (SBP) ≥140mmHg and/or diastolic blood pressure (DBP) ≥90mmHg
  Interventions: Procedure: Mobil-O-Graph PWA
- Group N: Normotensive group (Group N): Other non-hypertensive patients
  Interventions: Procedure: Mobil-O-Graph PWA

INTERVENTIONS:
Procedure: Mobil-O-Graph PWA — After resting in a quiet room preoperatively, blood pressure was measured on the right arm using an oscillometric method.

SUMMARY:
Hypertension is a disease with increasing and serious complications all over the world. In particular, the incidence of hypertension increases with advancing age. Secondary problems that can be caused by hypertension include peripheral vascular diseases, arteriosclerosis, increased risk of heart attack and stroke. It is a measurement of pulse wave velocity (PWV), a non-invasive indicator of arterial stiffness. It is known that sudden hemodynamic changes that occur during the induction of anesthesia cause undesirable intraoperative and postoperative complications. It is known that arterial stiffness, which is more common in elderly patients, causes orthostatic hypotension in particular. For this reason, more hemodynamic instability may be seen in the general anesthesia procedure in elderly patients with increased arterial stiffness.

In our study, we aimed to investigate whether the hemodynamic changes observed during anesthesia induction in hypertensive elderly patients, whom we think have a high pulse wave velocity, are different from normotensive patients.

ELIGIBILITY:
Inclusion Criteria:

* According to the American Society of Anesthesiologists (ASA), physical condition I-II,
* Elective otolaryngology surgery with endotracheal intubation planned
* Patients aged 50 and over

Exclusion Criteria:

* Hypersensitivity to drugs
* Difficult intubation history
* Diabetes mellitus receiving insulin therapy
* Chronic renal failure or end-stage renal disease
* Heart failure (left ventricular ejection fraction ≤30%)
* Valve disease (moderate to severe)
* Atrial fibrillation

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All Patients aged 50 and over
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Difference between hemodynamic values | Basal measurement before induction of anesthesia, then at 1-minute intervals until after endotracheal intubation
  The difference between the hemodynamic values measured preoperatively and during anesthesia induction was calculated. In addition, ≥20% decrease in preoperative hemodynamic value and/or systolic blood pressure ≤90 mmHg hypotension, ≥20% increased hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University Faculty of Medicine, Department of Anesthesiology and Reanimation, Aydin, Turkey (Türkiye)